CLINICAL TRIAL: NCT00803569
Title: Phase I Study of ALVAC(2)-NY-ESO-1(M)/TRICOM (VCP2292) in Patients With Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Carcinoma Whose Tumors Express NY-ESO-1 or LAGE-1 Antigen
Brief Title: Vaccine Therapy in Stage II, III, or IV Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Roswell Park Cancer Institute (Other); New York University Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUD2007-005; CDR0000628730 (Other: Ludwig)
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2022-10

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; fallopian tube cancer; peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — sargramostim

STUDY DESIGN:
Intervention Model Description: All patients received the same study treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALVAC(2)-NY-ESO-1(M)/TRICOM + GM-CSF (Experimental): Patients received SC injections with ALVAC(2)-NY-ESO-1(M)/TRICOM (0.5 mL) on Day 1 and the GM-CSF sargramostim (100 μg) on Days 1 through 4 in continuous 28-day cycles for up to 6 cycles.
  Interventions: Biological: ALVAC(2)-NY-ESO-1(M)/TRICOM vaccine; Biological: Sargramostim

INTERVENTIONS:
Biological: ALVAC(2)-NY-ESO-1(M)/TRICOM vaccine — The vaccine comprises the modified canary pox vector, ALVAC(2), inserted with the following genes: NYESO-1(M), TRICOM (LFA-3, ICAM-1, B7.1), vvE3L, vvK3L. The vaccine is administered at a dose of 0.5 mL SC.
Biological: Sargramostim — The GM-CSF sargramostim is administered at a dose of 100 μg SC.

SUMMARY:
This was a Phase 1, non-randomized, open-label, multicenter study of the ALVAC(2)-NY-ESO-1(M)/TRICOM vaccine administered with the granulocyte macrophage-colony stimulating factor (GM-CSF) sargramostim in patients with NY-ESO-1- or LAGE-1-positive epithelial ovarian, fallopian tube, or primary peritoneal cavity cancers who had completed standard therapy for primary or recurrent disease and would have normally entered a period of observation. The primary study objective was to determine the safety and tolerability of study vaccination, with secondary objectives including the determination of clinical and immunological responses.

DETAILED DESCRIPTION:
Patients received subcutaneous (SC) injections with 0.5 mL of ALVAC(2)-NY-ESO-1(M)/TRICOM on Day 1 and 100 μg of the GM-CSF sargramostim on Days 1 through 4 in continuous 28-day cycles for up to 6 cycles. No dose escalation of either vaccine component was permitted. Patients received study vaccinations until disease progression or unacceptable toxicity.

Safety was evaluated by continuous monitoring of adverse events (AEs), concomitant medications, and vital signs, as well as through hematology and chemistry laboratory testing and physical examinations. Efficacy was determined through tumor response evaluations, cancer antigen (CA)-125 levels, and cellular and humoral immune responses (i.e., NY-ESO-1-specific T cells, antibodies to NY-ESO-1 and ALVAC, and delayed-type hypersensitivity [DTH] testing).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented epithelial carcinoma arising in the ovary, fallopian tube or peritoneum, from stage II-IV at diagnosis, treated with initial surgery and chemotherapy with at least one platinum-based chemotherapy regimen.
2. Complete response to frontline therapy as evidenced by negative clinical examination, CA-125 tumor marker, and computed tomography (CT) scan. In addition, if second look surgery was performed (by laparoscopy or laparotomy), the result must have been either negative or microscopic positive. These patients would have normally entered a period of observation after standard management.
3. Patients with recurrent disease were eligible if they had completed surgery and/or chemotherapy for recurrent disease and would have normally entered a period of observation after completion of standard management. Eligible patients could have had asymptomatic residual measurable disease on physical examination and/or CT scan, and/or could have had an elevated CA-125 or could have been in complete clinical remission (defined as a serum CA-125 ≤ 35 IU/mL, CT scan without objective evidence of disease, and normal physical examination).
4. Tumor expression of 1) NY-ESO-1 by reverse transcription-polymerase chain reaction (RT-PCR) (preferably) or immunohistochemistry (IHC); or 2) LAGE-1 by RT-PCR. Patients whose primary surgery was performed outside the study site were pre-screened and required to release tissue sections or blocks to the study site in order to determine tumor expression of NY-ESO-1 by IHC.
5. Expected survival of at least 6 months.
6. Full recovery from surgery.
7. Karnofsky performance status of 70 or more.
8. Laboratory parameters for vital functions were required to be in the normal range. Laboratory abnormalities that were not clinically significant were generally permitted, except for the following laboratory parameters, which were required to be within the ranges specified:

   * neutrophil count: ≥ 1.5 × 10^9/L
   * lymphocyte count: ≥ 0.5 × 10^9/L
   * platelet count: ≥ 100 × 10^9/L
   * serum creatinine: ≤ 2 mg/dL
   * serum bilirubin (total): ≤ 2 mg/dL
   * hemoglobin: ≥ 10 g/dL
9. Have been informed of other treatment options.
10. Age ≥ 18 years.
11. Able and willing to give valid written informed consent.

Exclusion criteria:

1. Metastatic disease to the central nervous system for which other therapeutic options, including radiotherapy, may have been available.
2. Other serious illnesses (e.g., serious infections requiring antibiotics, bleeding disorders).
3. History of autoimmune disease (e.g., thyroiditis, lupus) except vitiligo.
4. Other malignancy within 3 years prior to entry into the study, except for treated non-melanoma skin cancer and cervical carcinoma in situ.
5. Known immunodeficiency or human immunodeficiency virus positivity.
6. Known allergy or history of life-threatening reaction to GM-CSF.
7. Known allergies to eggs, neomycin, and bovine products, determined by history.
8. History of severe allergic reactions to vaccines or unknown allergens.
9. Myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, chest pain or shortness of breath with activity, or other heart conditions being treated by a doctor.
10. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dosing of study agent.
11. Mental impairment that could have compromised the ability to give informed consent and comply with the requirements of the study.
12. Lack of availability for immunological and clinical follow-up assessment.
13. Previous NY-ESO-1 vaccine therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-11-14 (Actual); Primary Completion 2011-01-24 (Actual); Study Completion 2011-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kunle Odunsi, MD, PhD, Study Chair — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Withers HG, Matsuzaki J, Long M, Rosario SR, Chodon T, Tsuji T, Koya R, Yan L, Wang J, Keler T, Lele SB, Zsiros E, Lugade A, Hutson A, Blank S, Bhardwaj N, Shrikant P, Liu S, Odunsi K. mTOR inhibition modulates vaccine-induced immune responses to generate memory T cells in patients with solid tumors. J Immunother Cancer. 2025 Mar 25;13(3):e010408. doi: 10.1136/jitc-2024-010408. PMID 40132910

RESULTS

PARTICIPANT FLOW:
Groups:
- ALVAC(2)-NY-ESO-1(M)/TRICOM + GM-CSF: Patients received subcutaneous (SC) injections with ALVAC(2)-NY-ESO-1(M)/TRICOM (0.5 mL) on Day 1 and the granulocyte macrophage-colony stimulating factor (GM-CSF) sargramostim (100 μg) on Days 1 through 4 in continuous 28-day cycles for up to 6 cycles.
Period: Overall Study
Arm/Group | ALVAC(2)-NY-ESO-1(M)/TRICOM + GM-CSF
Started | 13
Completed | 9
Not Completed | 4
Not completed — Progressive Disease | 3
Not completed — Noncompliance | 1

BASELINE CHARACTERISTICS:
Population: All enrolled patients.
Arm/Group | ALVAC(2)-NY-ESO-1(M)/TRICOM + GM-CSF
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.7 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment-emergent Adverse Events
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0. Treatment-emergent adverse events (TEAEs) were reported based on clinical laboratory tests, physical examinations, and vital signs from pre-treatment through the study period.
Time Frame: Continuously for up to 26 weeks
Population: Patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ALVAC(2)-NY-ESO-1(M)/TRICOM + GM-CSF
Number analyzed (Participants) | 13
Participants
  Any TEAE | 12
  Maximum Grade 1 TEAE | 6
  Maximum Grade 2 TEAE | 6
  Treatment-related TEAE | 12
  SeriousTEAE | 0
  Death | 0
  TEAE Leading to Discontinuation | 0

2. Secondary Outcome: Number of Patients With Best Overall Tumor Response
Description: Tumor responses were evaluated using computed tomography and categorized according to the Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0) at baseline, at Week 12 (± 28 days), and at Week 24 (end of study). Per RECIST, target lesions are categorized as follows: Complete Response (CR): Disappearance of all target lesions [no evidence of disease]; Partial Response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD): small changes that do not meet above criteria.
Time Frame: Baseline and Weeks 12 and 24
Population: Patients with data available from at least 1 post-baseline response assessment. One patient discontinued the study prior to the Week 12 response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | ALVAC(2)-NY-ESO-1(M)/TRICOM + GM-CSF
Number analyzed (Participants) | 12
Participants
  No evidence of disease | 10
  Progressive disease | 2

3. Secondary Outcome: Median Progression-free Survival (PFS)
Description: PFS was calculated from the date of the first dose of study drug to the date of documented progression or death, whichever occurred first. Patients without disease progression or death had their observation time censored at the date of the last valid disease assessment. PFS was summarized using Kaplan-Meier product-limit estimators.
Time Frame: Baseline and up to approximately 24 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | ALVAC(2)-NY-ESO-1(M)/TRICOM + GM-CSF
Number analyzed (Participants) | 12
days | 167.5 [81 to 177]

4. Secondary Outcome: Median Cancer Antigen 25 (CA-125) Values on Study
Description: Blood samples were collected for CA-125 testing as a component of disease evaluations at Baseline and Weeks 8, 12, 16, 20, and 24 (end of study) or every 2 to 3 months on study according to standard institutional practice.
Time Frame: Baseline through Week 24
Population: as for outcome 2
Measure: Median (Full Range); unit: U/mL
Arm/Group | ALVAC(2)-NY-ESO-1(M)/TRICOM + GM-CSF
Number analyzed (Participants) | 12
U/mL
  Baseline | 8.6 [2.6 to 386.5]
  Week 8 | 9.7 [2.7 to 935.2]
  Week 12 | 7.4 [2.0 to 366.6]
  Week 16 | 9.4 [2.0 to 389.1]
  Week 20 | 9.0 [2.0 to 1181.1]
  Week 24 | 8.0 [2.8 to 1587.7]

5. Secondary Outcome: Number of Patients With NY-ESO-1 and LAGE-1 Antigen Positivity
Description: Blood samples were collected for measurement of NY-ESO-1 and LAGE-1 antigen positivity at Baseline and Weeks 4, 8 ,12, 16, 20, and 24 (end of study). Antibody testing was performed by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline through Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ALVAC(2)-NY-ESO-1(M)/TRICOM + GM-CSF
Number analyzed (Participants) | 12
Participants
  NY-ESO-1: BL positive, Post-BL positive | 2
  NY-ESO-1: BL negative, Post-BL positive | 10
  LAGE-1: BL positive, Post-BL positive | 1
  LAGE-1: BL negative, Post-BL positive | 3
  LAGE-1: BL negative, Post-BL negative | 2
  LAGE-1: Not evaluable | 6

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring between the signing of informed consent and the off-study date were documented, regardless of the causal relationship to study drug. AEs occurring after the first dose of study drug were considered treatment emergent (i.e., TEAEs). The AE reporting period for this study was up to 26 weeks.
Description: AE documentation included onset/resolution dates, severity using the NCI CTCAE (version 3.0), seriousness, study drug action taken, treatment, and outcome. In summaries, treatment-related AEs included those with a "possible", "probable", or "definite" relationship to study drug; preferred terms were counted only once per patient at the maximum reported grade.
Arm/Group | ALVAC(2)-NY-ESO-1(M)/TRICOM + GM-CSF
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 12/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALVAC(2)-NY-ESO-1(M)/TRICOM + GM-CSF (N=13)
Injection site pain (General disorders) | 8
Injection site erythema (General disorders) | 7
Injection site reaction (General disorders) | 6
Fatigue (General disorders) | 5
Injection site induration (General disorders) | 4
Injection site pruritus (General disorders) | 2
Injection site rash (General disorders) | 2
Chills (General disorders) | 1
Hypothermia (General disorders) | 1
Influenza-like illness (General disorders) | 1
Injection site nodule (General disorders) | 1
Injection site swelling (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Headache (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Vaginal infection (Infections and infestations) | 2
Acute sinusitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Palpitations (Cardiac disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Skin test positive (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1
Flushing (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less